CLINICAL TRIAL: NCT00057070
Title: Facilitating Implementation of the PHS Smoking Cessation Guidelines - RESET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Single Group | Masking: Single
Other Study IDs: TRX 01-080
Record Dates: First submitted 2003-03-27; First posted 2003-03-28 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2007-02

CONDITIONS: Smoking Cessation; Randomized Controlled Trial
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Other)
  Interventions: Procedure: Smoking cessation information, collection, and dissemination

INTERVENTIONS:
Procedure: Smoking cessation information, collection, and dissemination

SUMMARY:
The adverse impact of tobacco use on disease prevalence and health care costs is well documented. Hence, finding effective ways to reduce tobacco dependence is an essential component of improving the outcomes, quality and efficiency of VHA care. The U.S. Public Health Service (PHS) Smoking Cessation Clinical Practice Guideline provides specific recommendations for treating tobacco dependence. Despite their strong evidence base, however, these recommendations have not been fully integrated into clinical practice within the VHA. Recent data suggest that logistical difficulties associated with identifying and linking smokers with appropriate treatments may explain why the PHS Smoking Cessation Guideline has not been more broadly implemented.

DETAILED DESCRIPTION:
Background:

The adverse impact of tobacco use on disease prevalence and health care costs is well documented. Hence, finding effective ways to reduce tobacco dependence is an essential component of improving the outcomes, quality and efficiency of VHA care. The U.S. Public Health Service (PHS) Smoking Cessation Clinical Practice Guideline provides specific recommendations for treating tobacco dependence. Despite their strong evidence base, however, these recommendations have not been fully integrated into clinical practice within the VHA. Recent data suggest that logistical difficulties associated with identifying and linking smokers with appropriate treatments may explain why the PHS Smoking Cessation Guideline has not been more broadly implemented.

Objectives:

The primary objective of this study is to assess the effectiveness of an intervention for increasing the rate of tobacco dependence treatment in a population of smokers identified through the VA Pharmacy Benefits Management database. Secondary objectives of this study include (1) assessing the effect of the intervention on smoking cessation rates, and (2) developing options for overcoming potential barriers to broad implementation of the strategies.

Methods:

The effectiveness of the intervention will be evaluated using a multi-center, randomized, controlled trial. Veterans receiving a prescription for transdermal nicotine, nicotine gum, or bupropion for smoking cessation in the past year at one of the participating VHA facilities (as determined from Pharmacy Benefits Management records) will be eligible for the study. A total of 1,900 eligible veterans selected from five test sites will be randomly assigned to one of two groups: (1) patient phone call and tailored, computerized prompt to providers (intervention), or (2) usual care (control). The primary outcome is the proportion of patients receiving pharmacological or other smoking cessation treatment in the six month follow-up period, as assessed from VA pharmacy and outpatient data files. All patients will be recruited to a brief phone interview six months post-intervention to gather secondary outcome measure data related to smoking status, quit history, and use of smoking cessation assistance.

Status:

Data preparation and analysis.

ELIGIBILITY:
Inclusion Criteria:

Subjects must have received a prescription for a smoking cessation medication in 2002.

Exclusion Criteria:

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1900 (Estimated)
Dates: Start 2001-10; Study Completion 2003-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melissa R. Partin, PhD, Principal Investigator — Minneapolis VA Health Care System, Minneapolis, MN; Anne M. Joseph, MD MPH, Principal Investigator — Minneapolis VA Health Care System, Minneapolis, MN; Bonnie G. Steele, PhD RN, Principal Investigator — VA Puget Sound Health Care System Seattle Division, Seattle, WA
Locations (2):
- United States (2):
  - Minneapolis VA Health Care System, Minneapolis, MN, Minneapolis, Minnesota
  - VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington

REFERENCES:
- [Result] Partin MR, An LC, Nelson DB, Nugent S, Snyder A, Fu SS, Willenbring ML, Joseph AM. Randomized trial of an intervention to facilitate recycling for relapsed smokers. Am J Prev Med. 2006 Oct;31(4):293-9. doi: 10.1016/j.amepre.2006.06.021. Epub 2006 Aug 22. PMID 16979453
- [Result] Nelson DB, Partin MR, Fu SS, Joseph AM, An LC. Why assigning ongoing tobacco use is not necessarily a conservative approach to handling missing tobacco cessation outcomes. Nicotine Tob Res. 2009 Jan;11(1):77-83. doi: 10.1093/ntr/ntn013. Epub 2009 Jan 27. PMID 19246444
- [Result] Fu SS, Okuyemi KS, Partin MR, Ahluwalia JS, Nelson DB, Clothier BA, Joseph AM. Menthol cigarettes and smoking cessation during an aided quit attempt. Nicotine Tob Res. 2008 Mar;10(3):457-62. doi: 10.1080/14622200801901914. PMID 18324564
- [Result] Baines AD, Partin MR, Davern M, Rockwood TH. Mixed-mode administration reduced bias and enhanced poststratification adjustments in a health behavior survey. J Clin Epidemiol. 2007 Dec;60(12):1246-55. doi: 10.1016/j.jclinepi.2007.02.011. Epub 2007 Jun 29. PMID 17998079
- [Result] Fu SS, Partin MR, Snyder A, An LC, Nelson DB, Clothier B, Nugent S, Willenbring ML, Joseph AM. Promoting repeat tobacco dependence treatment: are relapsed smokers interested? Am J Manag Care. 2006 Apr;12(4):235-43. PMID 16610925